CLINICAL TRIAL: NCT05476601
Title: Culturally Adapted Manually Assisted Problem-Solving Intervention (CMAP) Plus CBT Based Motivational Interviewing for Self-Harm in Individuals with Substance Use Disorder in Pakistan: a Feasibility RCT
Brief Title: CMAP Plus Intervention for Self-harm in Individuals with Substance Use Disorder in Pakistan
Acronym: CMAP Plus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHAR M-CMAP Plus-003
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Self Harm; Substance-Related Disorders
MeSH Terms: conditions — Self-Injurious Behavior; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMAP Plus (Experimental): CMAP Plus is comprised of an existing culturally adapted manually assisted problem-solving intervention (CMAP) integrated with CBT based Motivational Interviewing (MICBT) called (CMAP Plus). The TAU of intervention group participants will be continued along with study intervention.
  Interventions: Behavioral: CMAP Plus
- TAU alone (No Intervention): This will be comprised of standard care they will be receiving from participating centres at recruitment sites. The standard care for individuals with SUD in Pakistan usually includes a 2-3-week detoxification programme, followed by 2 months of weekly 1:1 session along with some family sessions, followed by a period of support groups programmes.

INTERVENTIONS:
Behavioral: CMAP Plus — The CMAP Plus intervention will be delivered individually, weekly over a period of 12 weeks.
  Arms: CMAP Plus

SUMMARY:
Objectives:

To determine the feasibility and acceptability of the culturally adapted CMAP Plus CBT based Motivational Interviewing (MICBT) called CMAP Plus for self-harm in individuals with substance use disorder (SUD) in a feasibility randomised controlled trial.

To explore participants' experiences with CMAP Plus intervention.

Study design and setting:

The study will be a mixed-method feasibility randomised controlled trial of CMAP Plus as an intervention for Self-Harm in individuals with SUD in Pakistan. The study will be conducted in six major cities in Pakistan: Rawalpindi, Karachi, Peshawar, Hyderabad, Multan and Lahore.

Sample size:

A total of N=80 participants will be recruited from hospital settings and addiction rehabilitation centers in participating study sites.

DETAILED DESCRIPTION:
The study aims to determine the feasibility and acceptability of culturally Adapted Manually Assisted problem-solving intervention (CMAP) Plus MICBT for self-harm in individuals with SUD. The intervention will include specific strategies to identify and address obstacles in changing self-harm and drug-taking behaviour and offer ways to manage these difficulties from a cognitive-behavioural formulation. The intervention will also include CBT based mindfulness practice that involves learning to purposefully pay attention to ones inner and external experiences with an impartial non judging attitude. It can enable people to change the way they think and feel about their experiences, especially stressful experiences. The study will recruit a total of 80 participants from participating study sites, and prospective participants will be screened against eligibility criteria. Eligible consented participants will then be enrolled in the study. An independent statistician will randomise participants to one of the two study arms: 1) CMAP Plus (Intervention) along with Treatment As Usual (TAU); or 2) TAU alone. Each participant in the intervention arm will receive 12 individual, weekly sessions. Each session will take approximately 50-60 minutes. The sessions will be delivered at a place convenient to the participants. Trained therapists will deliver the intervention. The TAU will be comprised of standard care they will be receiving from participating centres at recruitment sites. Assessment measures will be administered before and after the intervention at 12th week. All assessments will be rater blind. After post-assessments at 12th week, a purposefully selected subset (stratified by age, gender, ethnicity, sexuality, religion, clinical and recovery scores) of participants will be invited for qualitative interviews to explore their experiences and satisfaction with the intervention. Participants will be interviewed within 1 week of their post-intervention by a trained qualitative researcher exploring their experience with CMAP Plus, the barriers and facilitators to engagement, and perceived benefits or negative experiences with the intervention. A sample of up to 15 interviews would be enough to achieve category saturation. On average, interviews will last for 60 minutes. The interview will be face-to-face or through telephone as an alternative to a face-to-face meeting to reduce the number of in-person meetings given the current context of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above.
* Individuals diagnosed with SUD on DSM-5 criteria of mental disorders.
* Having episodes of self-harm in last three months defined as a deliberate act to harm one's own body including but not limited to self-cutting, self-biting, self-poisoning, self-scratching, self-burning, self-hitting, pulling hair etc. assessed by deliberate self-harm inventory.
* Capable to give informed consent.
* Those who have completed detoxification process.

Exclusion Criteria:

* Participants with DSM-5 criteria of mental disorder other than SUD; due to a general medical condition or dementia, delirium, schizophrenia, bipolar disorder, personality disorders, learning disability or any other condition to the extent that engagement in the intervention would not be possible, e.g. communication difficulties.
* Unlikely to be available for outcome assessments (temporary residence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicator | From baseline to 12th week (at the end of intervention)
  The feasibility will be determined by collecting data on recruitment rates. The success criterion of feasibility will be to recruit > 50% of eligible participants. We will also record attrition (number of dropouts) and retention rate (the proportion of participants who complete the intervention period).
Acceptability indicator | From baseline to 12th week (at the end of intervention)
  The acceptability of intervention will be assessed using data on attendance. The criterion for acceptability is a mean attendance rate of >70% of sessions (at least 9 sessions).

SECONDARY OUTCOMES:
The deliberate self-harm inventory | From baseline to 12th week (at the end of intervention)
  The deliberate self-harm inventory is a 17-item, behaviorally based, a self- report questionnaire developed by the author to assess deliberate self-harm. This measure assesses various aspects of deliberate self-harm, including frequency, severity, duration, and type of self-harming behavior.
Beck scale for suicide ideation | From baseline to 12th week (at the end of intervention)
  A 19-item instrument for detecting and measuring the current intensity of patient-specific attitude, behavior, and specificity of patient thoughts to kill him/ herself during the past week.
Beck Hopelessness Scale | From baseline to 12th week (at the end of intervention)
  Beck hopelessness scale is to measure three aspects of hopelessness, feelings about the future, loss of motivation, and expectations to assess participants' feelings of hopelessness.
Severity of dependence scale | From baseline to 12th week (at the end of intervention)
  Severity of dependence scale contains five items, all of which are explicitly concerned with psychological components of dependence. These items are specifically concerned with impaired control over drug-taking and with preoccupation and anxieties about drug use. It can be used to measure the degree of dependence experienced by users of different types of drugs.
Depression Anxiety Stress Scale | From baseline to 12th week (at the end of intervention)
  Depression Anxiety Stress Scale is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety, and stress and consists of 7 items per subscale.
Euro-Qol-5 Dimensions scale | From baseline to 12th week (at the end of intervention)
  It's a standardised instrument to measure participants' health-related quality of life. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/ discomfort, and anxiety/ depression)
Client Service Receipt Inventory | From baseline to 12th week (at the end of intervention)
  Client Service Receipt Inventory will be used to get detailed description of the use of health services (including the informal sector faith healers/Imams) at 12th week follow up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, Principal Investigator — University of Manchester; Nasim Chaudhry, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Pakistan Recovery Oasis, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No